CLINICAL TRIAL: NCT01483131
Title: Effects of Strength Training Associated With Vascular Occlusion in Patients With Knee Osteoarthritis
Brief Title: Vascular Occlusion in Patients With Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vascular occlusion and OA
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low intensity resistance training (Experimental)
  Interventions: Other: Exercise training
- High intensity resistance training (Experimental)
  Interventions: Other: Exercise training
- Low intensity resistance training with vascular occlusion (Experimental)
  Interventions: Other: Resistance training with vascular occlusion

INTERVENTIONS:
Other: Exercise training — 12 weeks of resistance training twice a week.
  Arms: High intensity resistance training; Low intensity resistance training
Other: Resistance training with vascular occlusion — 12 weeks of resistance training with vascular occlusion twice a week
  Arms: Low intensity resistance training with vascular occlusion

SUMMARY:
Resistance exercise plus vascular occlusion may induce greater improvements in strength and muscle mass than resistance training alone. The investigators speculate this training strategy could be beneficial in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* BMI <39
* Knee Ostearthritis type II and III
* VAS (visual analogue scale) between 2 and 8

Exclusion Criteria:

* Hip osteoarthritis
* Use of NSAID

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
muscle strength | 12 weeks

SECONDARY OUTCOMES:
Quality of Life | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo -School of Medicine - Clinical Hospital, São Paulo, São Paulo, Brazil